CLINICAL TRIAL: NCT00831519
Title: Biochemical, Hematologic, and Inflammatory Effects of Diabetes on the Newborn
Brief Title: The Effect of Diabetes on the Newborn
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Principal Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: JB_6.08_1
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Macrosomial, GD
- Macrosomial, control

SUMMARY:
The aim of this study is to test and compare biochemical, hematological, and inflammatory factors in diabetic and healthy pregnant mothers and in their newborns.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who plan to deliver at Western Galilee Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
oxidative stress | Immediately after delivery by cesarean section
  New borns of diabetic mother may have oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital- Nahariya, Nahariya, Israel